CLINICAL TRIAL: NCT01858636
Title: Post-Market Study of the St. Jude Medical Angio-Seal™ V-Twist Integrated Platform (VIP) Vascular Closure Device
Acronym: SEAL PM
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL06818
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Vascular Closure
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Angio-Seal VIP Vascular Closure
  Interventions: Device: Angio-Seal VIP 6 French (6F) and 8 French (8F) devices

INTERVENTIONS:
Device: Angio-Seal VIP 6 French (6F) and 8 French (8F) devices — These devices are used for the vascular closure procedure

SUMMARY:
To characterize the clinical outcomes of Angio-Seal VIP with St. Jude Medical (SJM) collagen through the collection of device/procedure-related major vascular complications and time to hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires closure of femoral artery puncture resulting from arterial access procedure.
* Patient is ≥18 years of age.
* Patient is willing to provide written informed consent prior to study device use.
* Patient is willing and able to adhere to data collection and follow-up requirements.

Exclusion Criteria:

* Patient is participating in another clinical trial which has the potential to impact hemostasis.
* Patient has an active groin infection or systemic infection.
* Patient has undergone a vascular access procedure within the past 90 days.
* Patient has been previously enrolled in the study. (For patients undergoing multiple interventions within a timeframe of 90 days, only the initial procedure may constitute a study enrollment.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will be included in the study will be indicated for the procedure according to the Instructions for Use. Physicians should carefully select patients based on the IFU including a consideration of all warnings and precautions.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (4):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Institut für Diagnostiche und Interventionelle Radiologie, Frankfurt
  - Univ. des Saarlandes, Homburg
  - Herzzentrum Leipzig GMBH, Leipzig
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Medisch Spectrum Twente, Enschede

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Angio-Seal VIP Vascular Closure
Started | 235 (Subjects consented)
Device Deployment | 211
Completed | 207
Not Completed | 28
Not completed — No Device Deployment Attempted | 24
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subects with deployed devices
Groups:
- Angio-Seal VIP Vascular Closure: Angio-Seal VIP 6F and 8F devices: These devices are used for the vascular closure procedure
Arm/Group | Angio-Seal VIP Vascular Closure
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 145
Region of Enrollment [Number; unit: participants]
  Germany | 146
  Netherlands | 65

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Experiencing a Device or Procedure Related Major Vascular Complication
Description: Major vascular complications include:
  Access Site Complications:
  * Hematoma >10 cm in size requiring surgical or percutaneous intervention
  * Major bleeding requiring transfusion of ≥2 units of blood or requiring surgical or percutaneous intervention
  * Pain requiring a hospitalization extended for more than 24 hours or a new hospitalization, or percutaneous or surgical intervention
  * Infection requiring a hospitalization extended for more than 24 hours or a new hospitalization or treatment with IV antibiotics
  * A/V Fistula requiring medical intervention (percutaneous or surgical)
  * Pseudoaneurysm requiring medical intervention (percutaneous or surgical) b. Lower Limb Ischemia requiring surgical or medical intervention or resulting in permanent injury/impairment c. Retroperitoneal hemorrhage requiring intervention (percutaneous or surgical)
Time Frame: 30 days post procedure
Population: All subjects with device deployments.
Measure: Number (95% Confidence Interval); unit: % of subjects with MVCs
Groups:
- Deployed Subjects: Percentage of subjects who experienced a major vascular complication during 30-days post procedure.
Arm/Group | Deployed Subjects
Number analyzed (Participants) | 211
% of subjects with MVCs | 2.8 [NA to 5.5] — Per protocol, a one sided Fischer Exact test was performed. As a result, a lower confidence bound is not available.
Statistical Analysis 1: Comparison: Deployed Subjects; Ho: Pt ≥ 8% Ha: Pt < 8%, where Pt is the proportion of deployed subjects with a protocol-defined vascular complication; Test type: Superiority or Other; p = 0.0029, Fisher Exact; A one-sided Fisher's exact test was performed with a 95% upper confidence bound of 5.5%

2. Primary Outcome: The Percentage of Procedures Achieving Hemostasis Within 5 Minutes of Device Deployment.
Time Frame: within 5 minutes of device deployment
Measure: Number (95% Confidence Interval); unit: % of proc. w/hemostasis within 5 min
Units Other Than Participants: Procedures
Groups:
- Deployed Subjects: Subjects with Angio-Seal deployed
Arm/Group | Deployed Subjects
Number analyzed (Participants) | 211
Number analyzed (Procedures) | 213
% of proc. w/hemostasis within 5 min | 98.6 [96.4 to NA] — Per protocol, a one sided Fischer Exact test was performed. As a result an upper confidence bound is not available.
Statistical Analysis 1: Comparison: Deployed Subjects; Ho: St ≤ 90% Ha: St > 90%, where St is the proportion of deployed subjects achieving hemostasis within 5 minutes; Test type: Superiority or Other; p < 0.0001, Fisher Exact; A one-sided Fisher's exact test was performed with a 95% lower confidence bound of 96.4%

ADVERSE EVENTS:
Time Frame: 30 days
Description: A summary of all ADEs, Serious Adverse Events (SAEs), and non-serious vascular events
Groups:
- Deployed Subjects: Adverse Events (AEs) are provided for all subjects that underwent a study device deployment.
Arm/Group | Deployed Subjects
Serious Adverse Events (participants affected / at risk) | 34/211
Other Adverse Events (participants affected / at risk) | 31/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deployed Subjects (N=211)
Coronary Artery Disease (Cardiac disorders) | 4 (4)
VASC bleeding (Vascular disorders) | 4 (4)
VASC pseudoaneurysm (Vascular disorders) | 4 (4)
Vascular Hematoma (Vascular disorders) | 4 (4)
Aortic Valve Stenosis (Cardiac disorders) | 3 (3)
Bacterial Infection (Infections and infestations) | 3 (3) — Vascular Access Site Complication (VASC) Infections
Atrial Fibrillation (Cardiac disorders) | 2 (3)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Vascular Disection (Vascular disorders) | 1 (1) — Coronary Site - Not Access Site
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (2)
Angina Pectoris (Cardiac disorders) | 1 (1)
Decreased Left Ventricular Function (Cardiac disorders) | 1 (1)
Elective Cardiac Surgery (Cardiac disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Intracerebral Hemorrhage (Vascular disorders) | 1 (1)
Ischemic Stroke (Vascular disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1)
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deployed Subjects (N=211)
VASC bruise (Vascular disorders) | 17 (17)
VASC hematoma (Vascular disorders) | 8 (9)
VASC bleeding (Vascular disorders) | 5 (5)
VASC pain (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No